CLINICAL TRIAL: NCT00462319
Title: Evaluation of Standardized Management of Knee Arthritis Patients
Brief Title: ARTIST: ARThrose Intervention STandardisée
Acronym: ARTIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 2004/07
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Education, weight reduction and physical exercise

SUMMARY:
International recommendations (ACR,EULAR) emphasize physical exercise and weight loss for patients suffering from knee osteoarthritis. Nevertheless, number of patients receiving advices for these 2 points still low. This study evaluates the impact of a standardized medical intervention (patient education, weight reduction and physical exercise) in knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic and ambulatory patients
* suffering from knee osteoarthritis (ACR criteria)
* 25<BMI<35
* signed informed consent

Exclusion Criteria:

* need to surgery within 6 next months
* co-morbidity

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05

PRIMARY OUTCOMES:
Weight
Physical Exercise in Leisure

CONTACTS AND LOCATIONS:
Overall Officials: René Marc FLIPO, Principal Investigator — Hôpital Salengro - Lille, France
Locations (1):
- Paris, France

REFERENCES:
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] Messier SP, Gutekunst DJ, Davis C, DeVita P. Weight loss reduces knee-joint loads in overweight and obese older adults with knee osteoarthritis. Arthritis Rheum. 2005 Jul;52(7):2026-32. doi: 10.1002/art.21139. PMID 15986358
- [Derived] Ravaud P, Flipo RM, Boutron I, Roy C, Mahmoudi A, Giraudeau B, Pham T. ARTIST (osteoarthritis intervention standardized) study of standardised consultation versus usual care for patients with osteoarthritis of the knee in primary care in France: pragmatic randomised controlled trial. BMJ. 2009 Feb 23;338:b421. doi: 10.1136/bmj.b421. PMID 19237406